CLINICAL TRIAL: NCT02789228
Title: Research Study Utilizing Expanded Multi-antigen Specific Lymphocytes for the Treatment of Solid Tumors
Acronym: REST
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, HMeany, Associate Professor and Hematology-Oncology Fellowship Director, Children's National Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7497
Record Dates: First submitted 2016-05-24; First posted 2016-06-02 (Estimated); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Group A includes patients who have undergone an allogeneic hematopoietic stem cell transplant (HSCT) as part of their prior therapy.
  Group A patients (post allogeneic HSCT): TAA-T will be infused any time after neutrophil engraftment post-HSCT or day 30, whichever comes first.
  Interventions: Biological: Tumor associated antigen lymphocytes (TAA-CTL)
- Group B (Experimental): Group B includes patients who have undergone conventional (standard) therapy which does not include an allogeneic HSCT. Within group B, a cohort of patients with relapsed or refractory Wilms tumor will be enrolled and receive a lymphodepleting chemotherapy regimen followed by TAA-T.
  Group B patients (no prior allogeneic HSCT): TAA-T will be infused any time >1 week after completing most recent course of conventional (non-investigational) therapy for their disease. Patients receiving lymphodepletion will be >2 weeks from most recent course of conventional therapy and have nadired and recovered before beginning protocol therapy.
  Interventions: Biological: Tumor associated antigen lymphocytes (TAA-CTL)

INTERVENTIONS:
Biological: Tumor associated antigen lymphocytes (TAA-CTL) — This protocol is designed as a phase I dose-escalation study. In each treatment group (A and B), patients will be enrolled to one of the following TAA-T dose levels:
  Dose Level One: 1 x 107 cells/m2 Dose Level Two: 2 x 107 cells/m2 Dose Level Three: 4 x 107 cells/m2

SUMMARY:
Patients with high-risk solid tumors, those that are refractory to standard up front therapy or relapse after completion of therapy, have a very poor prognosis despite attempts to induce remission with salvage regimen. Novel therapies are critical for this patient population with high-risk cancer.

The ability of tumors to be recognized and lysed by the immune system offers a unique opportunity to aid in tumor eradication by expanding and activating these anti-tumor cells. Through this ability to harness sophisticated and specific immunotherapy, residual or relapsed disease that is resistant to chemotherapy and/or radiotherapy could be eradicated. Prior studies have suggested both safety of expanded specific T cells and efficacy in the setting of melanoma, lymphoma or viral eradication. While this therapy has previously been limited by the versatility of the tumor to down-regulate antigens and evade a single immune-target, the use of multi-antigen specific T cells may permit better and more durable anti-tumor immunity. Thus, the investigators propose to infuse these specific multi-antigen anti-tumor T lymphocytes into patients with high risk solid tumors. This trial will be conducted to demonstrate safety of these cells and generate efficacy and biology data that may be important for future studies that may enhance tumor immunotherapy.

DETAILED DESCRIPTION:
This protocol is designed as a phase I dose-escalation study. In each treatment group (A and B), patients will be enrolled to one of the following TAA-CTL dose levels:

Dose Level One: 1 x 107 cells/m2 Dose Level Two: 2 x 107 cells/m2 Dose Level Three: 4 x 107 cells/m2

Patients will receive cells due to the presence of refractory disease and/or high risk for disease relapse and/or residual detectable disease following HSCT or conventional therapy at the time of the infusion. Group A and Group B patients will use the dose escalation strategy described above. Ideally, patients should not receive other systemic antineoplastic agents for at least 45 days after the infusion of TAA- CTL (for purposes of evaluation), although such treatment may be added if deemed critical for patient care by the attending physician.

Two to four patients will be enrolled at each dose level until the maximum tolerated dose (MTD) is determined at which point to ensure safety a total 8 patients will be treated at the MTD. Each patient will receive at least one TAA-CTL infusion and may receive a maximum of 8 doses total. Dose escalation will occur once at least 2 patients have completed the 45 day follow up period following their first TAA-CTL infusion. The first and second doses will be administered 45 days apart then additional doses will be spaced every 28 days. The expected volume of each infusion is 1 to 10 cc.

Expansion cohorts of Group B patients with Wilms tumor, neuroblastoma, rhabdomyosarcoma, adenocarcinoma and esophageal cancer will be permitted to enroll up to 6 additional patients in each disease group, to be treated at the MTD.

Within group B, a cohort of patients with relapsed or refractory Wilms tumor will be enrolled and receive a lymphodepleting chemotherapy regimen followed by TAA-T.

If patients with measurable or evaluable disease have a response of stable disease or better by RECIST criteria at the day 28 evaluation after dose 2 or subsequent evaluations they are eligible to receive up to 6 additional doses of CTLs at 28 day intervals. Each subsequent doseis expected to be at the enrollment dose level (i.e. no subsequent dose escalation). Following dose 1, if a patient's T cell supply is insufficient for subsequent doses at the enrollment dose level, further treatments may be administered at a lower dose level at the treating physician's discretion.

ELIGIBILITY:
Inclusion Criteria:

Recipient procurement inclusion criteria

* Diagnosis of high-risk solid tumors: Ewing sarcoma, Wilms tumor, neuroblastoma, rhabdomyosarcoma, soft tissue sarcomas, osteosarcoma, adenocarcinoma, and esophageal carcinoma and renal cell carcinoma.
* Refractory disease, residual detectable disease following conventional therapy or relapsed disease.
* 6 months to 60 years of age at enrollment.*
* Karnofsky/Lansky score of ≥ 50%.*
* Absolute neutrophil count (ANC) greater than 500/µL. *
* Absolute lymphocyte count (ALC) greater than 1000/µL.*
* Bilirubin ≤ 2.5 mg/dL. *
* Aspartate aminotransferase (AST)/ Alanine transaminase (ALT) ≤ 5x the upper limit of normal for age. *
* Serum creatinine < 1.0 mg/dL or 2 x the upper limit of normal for age (whichever is higher).*
* Pulse oximetry of > 90% on room air.*
* Agree to use contraceptive measures during study protocol participation (when age appropriate).*
* LVEF > 50% or LVSF > 27 % if history of total body irradiation (TBI).
* Patient or parent/guardian capable of providing informed consent.

Exclusion Criteria:

Recipient Procurement exclusion criteria

* Patients with uncontrolled infections
* Patients with active HIV
* Current evidence of GVHD > grade 2 or chronic GVHD manifestations: bronchiolitis obliterans syndrome, sclerotic GVHD, or serositis.
* Pregnant or lactating females
* Prior immunotherapy with an investigational agent within the last 28 days prior to procurement

Recipient Inclusion to administer cells:

* Steroids less than 0.5 mg/kg/day prednisone (or equivalent).
* Karnofsky/Lansky score of ≥ 50% %.
* Bilirubin ≤ 2.5 mg/dL.
* AST/ALT ≤ 5x the upper limit of normal for age.
* Serum creatinine < 1.0 mg/dL or 2x the upper limit of normal for age (whichever is higher).
* Pulse oximetry of > 90% on room air.
* Patients receiving lymphodepleting chemotherapy must have:

ANC >750 /uL Platelet count >75,000 /uL

Recipient Exclusion to administer cells:

* Patients with uncontrolled infections
* Patients who received ATG, Campath, or other T cell immunosuppressive monoclonal antibodies within 28 days prior to TAA-T cell infusion
* Acute GVHD > grade 2 or chronic GVHD manifestations: bronchiolitis obliterans syndrome, sclerotic GVHD, or serositis
* Pregnant or lactating females

Ages: 6 Months to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Product-Emergent Adverse Events | Within 45 days of the last dose of TAA-CT of first infusion and 28 days after the final TAA CTL dose
  Primary endpoint of the study is defined grade ≥3 infusion-related adverse event occurring within 45 days of the last TAA-CTL dose, grade ≥4 non-hematologic adverse event occurring within 45 days of the last TAA-CTL dose and that are not due to the patient's underlying malignancy or pre-existing co-morbidities or grade ≥3 acute GVHD occurring within 45 days of the last TAA-CTL dose, or any unexpected toxicity of any grade attributed to the infusion of TAA-CTL occurring within 45 days of the last TAA-CTL dose. Toxicities will be defined by the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 4.03

SECONDARY OUTCOMES:
Tumor associated antigen lymphocytes (TAA-CTL) responses | 1 year
  o determine the number of patients who respond to tumor associated antigen lymphocytes (TAA-CTL)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hont AB, Cruz CR, Ulrey R, O'Brien B, Stanojevic M, Datar A, Albihani S, Saunders D, Hanajiri R, Panchapakesan K, Darko S, Banerjee P, Fortiz MF, Hoq F, Lang H, Wang Y, Hanley PJ, Dome JS, Bollard CM, Meany HJ. Immunotherapy of Relapsed and Refractory Solid Tumors With Ex Vivo Expanded Multi-Tumor Associated Antigen Specific Cytotoxic T Lymphocytes: A Phase I Study. J Clin Oncol. 2019 Sep 10;37(26):2349-2359. doi: 10.1200/JCO.19.00177. Epub 2019 Jul 29. PMID 31356143